CLINICAL TRIAL: NCT04170088
Title: Comparison of Efficacy of Tranexamic Acid Mesotherapy Versus 0.9% Normal Saline for Melasma; a Split Face Study in Tertiary Care Hospital of Karachi
Brief Title: Comparison of Efficacy of Tranexamic Acid Mesotherapy Versus 0.9% Normal Saline for Melasma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr Sana Kaleem, Department of Dermatology, SKaleem, FCPS II Postgraduate Trainee, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: F.2-81/2018-GENL/2522/JPMC; sana.dec04@hotmail.com (Registry Identifier: JinnaH Postgraduate Medical Centre)
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-11

CONDITIONS: Effect of Drugs; Adverse Effects of Medical Drugs
Keywords: Melasma; Tranexamic acid; Mesotherapy
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: individual patients were selected in study . To control over confounding factors two sides of same patient were used parallel for intradermal injection ( Mesotherapy) of tranexamic acid and with normal saline
Who Masked: Participant, Care Provider
Masking Description: Participant do not know about the split face study. Their one side was injected by tranexamic acid diluted in normal saline while other side was injected with simple normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Experimental): Left side of face of each participant was selected for intradermal Tranexamic acid injections.
  generic name : Tranexamic acid Dose : 4mg / ml tranexamc acid diluted with 0.9 % normal saline Frequency : every 2 weekly total 6 doses. Duration : 6 months
  Interventions: Drug: Tranexamic Acid; Drug: 0.9% Normal Saline
- 0.9% Normal saline (Experimental): Right side of face of each participant was selected for intradermal normal saline injections generic name : Normal Saline Dose : 0.9 % Normal Saline Dose : Frequency : every 2 weekly total 6 doses. Duration : 6 months
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid intradermal injections were used for treatment of melasma
  Other Names: Normal saline
  Arms: Tranexamic acid
Drug: 0.9% Normal Saline — Normal saline used for comparision of efficacy of tranexamic acid

SUMMARY:
It is a randomized controlled trial in which investigators determine the efficacy of tranexamic acid (TA) by mesotherapy in comparison to normal saline on participants having Melasma.

DETAILED DESCRIPTION:
In this prospective single blind split face controlled trial.Total 30 patients referred to Dermatology Ward were selected. At first, patients were examined under wood lamp for determination of melasma type (epidermal, dermal). Then, patients underwent Tranexamic acid microinjections with a concentration of TA 4 mg/ml with 0.9 % normal saline on their left half of the face and only 0.9%normal saline on their right half of the face, with mesotherapy technique. This procedure was done total of six times with 2-week intervals. Participants were assessed by Hemi Modified Melasma Area and Severity Scoring (mMASI) at start and end of the study for each half of face. Statistical Package for Social Sciences (SPSS) , version 23 was used for analysis. P value < 0.01 was taken significant.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 18 to 55 years
* bilateral symmetrical mild to severe melasma

Exclusion Criteria:

* pregnancy and lactation
* history of taken any topical treatment for melasma in previous 1 month
* history of bleeding disorders
* concomitant use of anticoagulants,
* any known drug allergy especially to the study drug,
* having associated medical illnesses.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in HEMI-Modified Melasma Area and Severity Index (mMASI) | 10 months
  Calculation of Hemi mMASI score is performed by rating darkness and area of involvement of 3 areas of the each half of face. These figures are then inserted into an equation, resulting in the final Hemi mMASI score for both halves of face. Equation : forehead (0.15×D×A) + malar ( 0.30×D×A) + chin ( 0.05×D×A) The mean value of the data obtained from each half of the face was calculated and the mean percentage change was compared. Hemi-MASI score was used because of the study design of split-face, and it was calculated based on the percentage of the involved area Improvement was considered when there was reduction in mean hemi modified MASI score at both sides of face. Higher score was considered as worse and low score was considered as good in improvement of melasma.
  At each follow-up visit, adverse events were also evaluated. Patients were asked to reports side effects such as erythema, burning, swelling, and change in menstrual cycle during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: rabia ghafoor, FCPS, Study Director — Assistant Profesor
Locations (1):
- Jinnah potgraduate Medical Centre ( JINNAH HOPITAL), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ogbechie-Godec OA, Elbuluk N. Melasma: an Up-to-Date Comprehensive Review. Dermatol Ther (Heidelb). 2017 Sep;7(3):305-318. doi: 10.1007/s13555-017-0194-1. Epub 2017 Jul 19. PMID 28726212
- [Result] Handel AC, Miot LD, Miot HA. Melasma: a clinical and epidemiological review. An Bras Dermatol. 2014 Sep-Oct;89(5):771-82. doi: 10.1590/abd1806-4841.20143063. PMID 25184917